CLINICAL TRIAL: NCT02926703
Title: Lactate Compared to Creatine Kinase as Diagnostic Marker in Generalized Epileptic Seizure
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: Laktat-2016; EK 267/15 (Other: local ethics committee)
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-09

CONDITIONS: Seizure; Syncope
Keywords: seizure; lactate; creatine kinase
MeSH Terms: conditions — Seizures; Syncope | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2-5 ml blood sample for the measurements of serum lactate and creatine kinase concentrations
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GTCS patients: Patients with generalized tonic-clonic seizures (GTCS) and whose serum lactate and creatine kinase (CK) concentrations in blood samples had been measured within 2 hours after the event. In a subgroup of patients follow up blood samples were taken at 10 to 48 hours after the seizure to allow longitudinal the comparison of both markers
  Interventions: Other: Serum lactate and CK concentrations in blood samples
- Syncope patients: Patients with syncope and whose serum lactate and CK concentrations in blood samples had been measured within 2 hours after the event. In a subgroup of patients follow up blood samples were taken at 10 to 48 hours after the seizure to allow longitudinal the comparison of both markers.
  Interventions: Other: Serum lactate and CK concentrations in blood samples

INTERVENTIONS:
Other: Serum lactate and CK concentrations in blood samples — Serum lactate and CK concentrations in blood samples were measured routinely at admission

SUMMARY:
The investigators compared the feasibility of serum creatine kinase and serum lactate concentration as diagnostic markers to distinguish between generalized tonic-clonic seizures (GTCS) and syncopes in clinical settings that require fast-action treatment, such as in the emergency departments.

DETAILED DESCRIPTION:
The patients of this prospective study were selected from a sample of patients who were admitted to the emergency room of the University Hospital RWTH Aachen with an unclear impairment of consciousness. Only patients who later on were diagnosed as having experienced a GTCS or a syncope and whose serum lactate concentrations had been measured within 2 hours after the event were enrolled in the study. The investigators compared the specificity and sensitivity of the serum lactate concentrations at admission with the CK concentration at admission and the CK follow-up taken 10 to 48 hours after the event.

The values at admission were compared between patients from whom a blood sample was collected within 60 minutes after the event, and those from whom a blood sample was collected within 61-120 minutes after the event.

The comparison of initial lactate concentrations at admission with CK levels 10 - 48 hours later could only be performed on part of the patient collective because the other patients were already discharged at this time-point and could therefore not be included.

The initial blood samples were taken at patient arrival in the emergency room. The follow up was performed during the inpatient stay.

Serum lactate and CK concentrations between patient groups were statistically compared with a Mann-Whitney-U test. We defined cut-off values and their sensitivity and specificity by Receiver Operating Characteristic (ROC) analysis.

ELIGIBILITY:
Inclusion Criteria:

Patients with generalized tonic-clonic seizures and syncopes and whose blood samples were taken within 2 hours after the event

18 years or older

Observed seizure

Time of the event before admission was known

Diagnosis of an epileptic seizure or syncope had been entered in the final discharge report

Exclusion Criteria:

Prisoner

Age < 18 years old

Competing explanations for serum lactate or CK elevation e.g. shock or trauma

Lack of capacity for consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department patients
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Comparison of the first measurements of serum lactate and creatine kinase concentrations in blood samples between patients admitted with either a generalized tonic-clonic seizure or a syncope | 2 hours

SECONDARY OUTCOMES:
Comparison of the serum lactate concentrations at admission with the CK follow-up taken 10 to 48 hours after the event | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Dafotakis, Dr., Study Director — Department of Neurology, University Hospital RWTH Aachen, Germany
Locations (1):
- Department of Neurology/Emergency department, University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matz O, Zdebik C, Zechbauer S, Bundgens L, Litmathe J, Willmes K, Schulz JB, Dafotakis M. Lactate as a diagnostic marker in transient loss of consciousness. Seizure. 2016 Aug;40:71-5. doi: 10.1016/j.seizure.2016.06.014. Epub 2016 Jun 23. PMID 27367837